CLINICAL TRIAL: NCT02161588
Title: A Multiple Dose, Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Assess the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Oral Semaglutide in Healthy Male Japanese and Caucasian Subjects
Brief Title: A Trial to Assess the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Oral Semaglutide in Healthy Male Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4140; U1111-1148-4141 (Other: WHO); JapicCTI-142572 (Other: JAPIC)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Once-daily oral administration as tablets. The dose level of oral semaglutide used in the 'Dose escalation period', 'Treatment period 1', 'Treatment period 2' and 'Treatment period 3' will be 5, 10, 20 and 40 mg per day, respectively.
  Arms: Semaglutide
Drug: placebo — Once-daily oral administration as tablets.
  Arms: Placebo

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body), pharmacodynamics (the effect of the investigated drug on the body), safety and tolerability of oral semaglutide in healthy male Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Japanese and Caucasian subjects
* Age between 20 and 55 years (both inclusive) at time of signing informed consent
* Body weight of above or equal to 54.0 kg
* Body mass index (BMI) between 20.0 and 25.0 kg/m^2 (both inclusive)
* Glycosylated haemoglobin A1c (HbA1c) below or equal to 6.0%

Exclusion Criteria:

* Presence or history of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, GI (gastrointestinal), endocrine, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders, as judged by the investigator. Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Smoking of more than 5 cigarettes (including nicotine substitute products), or the equivalent, per day or unwilling to refrain from smoking whenever required for the trial procedure
* Use of prescription drugs within 3 weeks or 5 times the half-life, whichever is longer, prior to Visit 2 (Day 1), non-prescription drugs within 1 week prior to Visit 2 (Day 1). The use of vitamins and minerals, and the occasional use of paracetamol (acetaminophen) or acetylsalicylic acid are permitted
* Any blood drawn in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening
* Previous GI surgery such as invasive and corrective procedures involving the oesophagus, stomach, duodenum, gallbladder (e.g., cholecystectomy), pancreas or intestinal resections. Exempt are subjects that underwent uncomplicated surgical and diagnostic procedures such as appendectomy, hernia surgery, polypectomy, biopsies, as wells as colonic and gastric endoscopy

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration-time curve | During a dosing interval (0-24 hours) at steady state

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | During a dosing interval (0-24 hours) at steady state
Number of treatment emergent adverse events (TEAEs) recorded | From the time of first dosing (Day 1) until completion of the follow-up visit (Days 119-126)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com